CLINICAL TRIAL: NCT00218036
Title: Pharmacotherapy Dosing Regimen in Cocaine and Opiate Dependent Individuals
Brief Title: Pharmacotherapy Dosing Regimen in Cocaine and Opiate Dependent Individuals - 8
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution, end of funding, clinic relocation, recruitment issues
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Texas (Other)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psy, Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-09262-8; P50DA009262-08 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Cocaine Abuse; Opiate Dependence
Keywords: Cocaine Abuse; Opiate Abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Modafinil; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Modafinil 200mg / Methadone Maintenance (1.2mg/kg)
  Interventions: Drug: Modafinil 200mg
- 2 (Experimental): Modafinil 400mg/ Methadone Maintenance (1.2mg/kg)
  Interventions: Drug: Modafinil 400mg
- 3 (Experimental): Citalopram 20/ Methadone Maintenance 1.2mg/kg
  Interventions: Drug: Citalopram 20mg
- 4 (Experimental): Citalopram 40/ Methadone Maintenance 1.2 mg/kg
  Interventions: Drug: Citalopram 40mg
- 5 (Placebo Comparator): Placebo given to methadone-maintained subjects (1.2mg/kg) for the duration of the 12-week study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil 200mg — 10 day medication run-up to Modafinil 200mg while subject is methadone maintained at 1/2 mg/kg. On full dose for 12 weeks and then titrated down for 10 days.
  Arms: 1
Drug: Modafinil 400mg — 10 day medication run-up to 400mg of Modafinil while subject is methadone maintained at 1.2 mg/kg. On full dose for 12 weeks and then titrated down for 10 days.
  Arms: 2
Drug: Citalopram 20mg — 10 day run-up to Citalopram 20mg while subject is methadone maintained at 1.2mg/kg. On full dose for 12 weeks and then titrated down for 10 days.
  Arms: 3
Drug: Citalopram 40mg — 10 day medication run-up to Citalopram 40 mg while subjects are methadone maintained (1.2 mg/kg). On full dose for 12 weeks and then titrated down for 10 days.
  Arms: 4
Drug: Placebo — Placebo while patient is methadone maintained on standard dose of 1.2 mg/kg
  Arms: 5

SUMMARY:
The purpose of this study is to examine two medications, modafinil and citalopram, in the treatment of cocaine dependent individuals who are maintained on methadone.

DETAILED DESCRIPTION:
This is a 24-week, randomized, double-blind, placebo-controlled study examining two doses of modafinil (200 and 400 mg) and citalopram (20 and 40 mg) in the treatment of methadone maintained cocaine dependent individuals.

Participants will first be given methadone to determine its tolerated and effective doses. Most participants will be able to reach a stable dose of methadone within 7 to 10 days of methadone initiation. When 80% of the projected dose of methadone has been achieved, participants will begin the medication regimen of modafinil or citalopram. Modafinil will be given over a 7-day period. Dosing of modafinil will begin at 200 mg and, depending on the individual, may increase to 400 mg. Citalopram will be given in increasing doses, starting at 20 mg and increasing to 40mg.

ELIGIBILITY:
Inclusion Criteria:

* Meets cocaine abuse and dependence criteria (as determined by the SCID)
* Meets opiate dependence criteria (as determined by the SCID)
* In good general physical and psychiatric health (except for possible acute drug use related problems)

Exclusion Criteria:

* Meets diagnostic criteria for other psychiatric disorders, including other forms of drug dependence (other than nicotine)
* Current cardiovascular disease (as determined by an electrocardiogram)
* Circumstances will not allow for completion of study (on probation or parole)
* Ethical constraints of supervision do not allow confidentiality (on probation or parole)

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy M Schmitz, PhD, Principal Investigator — University of Texas; F. Gerard Moeller, M.D., Study Chair — University of Texas Medical School at Houston
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 54 were enrolled, but only 51 were randomized and started the study.
Groups:
- Modafinil 200mg/Methadone Maintenance (1.2mg/kg): 10 day medication run-up to Modafinil 200mg while subject is methadone maintained at 1.2 mg/kg. On full dose for 12 weeks and then titrated down for 10 days.
- Modafinil 400mg/Methadone Maintenance (1.2mg/kg): 10 day medication run-up to 400mg of Modafinil while subject is methadone maintained at 1.2 mg/kg. On full dose for 12 weeks and then titrated down for 10 days.
- Citalopram 20mg/Methadone Maintenance (1.2mg/kg): 10 day run-up to Citalopram 20mg while subject is methadone maintained at 1.2mg/kg. On full dose for 12 weeks and then titrated down for 10 days.
- Citalopram 40mg/Methadone Maintenance (1.2mg/kg): 10 day medication run-up to Citalopram 40 mg while subjects are methadone maintained (1.2 mg/kg). On full dose for 12 weeks and then titrated down for 10 days.
- Placebo/Methadone Maintenance (1.2mg/kg): Placebo while patient is methadone maintained on standard dose of 1.2 mg/kg
Period: Overall Study
Arm/Group | Modafinil 200mg/Methadone Maintenance (1.2mg/kg) | Modafinil 400mg/Methadone Maintenance (1.2mg/kg) | Citalopram 20mg/Methadone Maintenance (1.2mg/kg) | Citalopram 40mg/Methadone Maintenance (1.2mg/kg) | Placebo/Methadone Maintenance (1.2mg/kg)
Started | 11 | 6 | 13 | 12 | 9
Completed | 6 | 3 | 5 | 6 | 3
Not Completed | 5 | 3 | 8 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil 200mg/Methadone Maintenance (1.2mg/kg) | Modafinil 400mg/Methadone Maintenance (1.2mg/kg) | Citalopram 20mg/Methadone Maintenance (1.2mg/kg) | Citalopram 40mg/Methadone Maintenance (1.2mg/kg) | Placebo/Methadone Maintenance (1.2mg/kg) | Total
Number analyzed (Participants) | 11 | 6 | 13 | 12 | 9 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.364 (11.474) | 40.333 (8.335) | 38.769 (7.350) | 36.500 (9.050) | 36.556 (7.618) | 37.510 (8.941)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 4 | 3 | 15
  Male | 8 | 5 | 9 | 8 | 6 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 6 | 13 | 12 | 9 | 51

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Abstinence From Cocaine
Time Frame: 12 weeks of treatment
Population: The trial was terminated when the PI of the study left the institution. Collected data was stored in a database management system that has since become obsolete and is no longer accessible by current database programs.
Arm/Group | Modafinil 200mg/Methadone Maintenance (1.2mg/kg) | Modafinil 400mg/Methadone Maintenance (1.2mg/kg) | Citalopram 20mg/Methadone Maintenance (1.2mg/kg) | Citalopram 40mg/Methadone Maintenance (1.2mg/kg) | Placebo/Methadone Maintenance (1.2mg/kg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Retention
Time Frame: 12 weeks of treatment
Population: as for outcome 1
Arm/Group | Modafinil 200mg/Methadone Maintenance (1.2mg/kg) | Modafinil 400mg/Methadone Maintenance (1.2mg/kg) | Citalopram 20mg/Methadone Maintenance (1.2mg/kg) | Citalopram 40mg/Methadone Maintenance (1.2mg/kg) | Placebo/Methadone Maintenance (1.2mg/kg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Medication Compliance
Time Frame: 12 weeks of treatment
Population: as for outcome 1
Arm/Group | Modafinil 200mg/Methadone Maintenance (1.2mg/kg) | Modafinil 400mg/Methadone Maintenance (1.2mg/kg) | Citalopram 20mg/Methadone Maintenance (1.2mg/kg) | Citalopram 40mg/Methadone Maintenance (1.2mg/kg) | Placebo/Methadone Maintenance (1.2mg/kg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The trial was terminated when the PI of the study left the institution. Collected data was stored in a database management system that has since become obsolete and is no longer accessible by current database programs.
Arm/Group | Modafinil 200mg/Methadone Maintenance (1.2mg/kg) | Modafinil 400mg/Methadone Maintenance (1.2mg/kg) | Citalopram 20mg/Methadone Maintenance (1.2mg/kg) | Citalopram 40mg/Methadone Maintenance (1.2mg/kg) | Placebo/Methadone Maintenance (1.2mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Difficulty recruiting and lower than desired sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No